# Effekt på QTc-tid av bytte fra (R,S)-metadon til (R)-metadon hos LAR-pasienter med kjent lang QTc-tid

**Innledning** Hovedhensikten med studien er å undersøke om en konvertering fra (R,S)-metadon og R-metadon kan normalisere QTc-tid hos risikopasienter.

Pasienter med kongenital eller ervervet lang QTc-tid kan risikere utvikling av potensielt alvorlige arytmier. En konvertering fra (R,S)-metadon og (R)-metadon kan imidlertid være et verdifult bidrag, i sær til pasienter som verken ønsker å redusere sin daglige metadondose eller å skifte til buprenorfin.

**Nøkkelord:** Substitusjonsbehandling, metadon, LAR, MMT, OMT, EKG, elektrokardiogram, kiral metadon, (R,S)-metadon, racemisk metadon, R-metadon, S-metadon, hjertearytmi, forlenget QTc-tid

Bakgrunn: Metadon ble utviklet av tyske forskere i 1937 som erstatter for morfin i smertebehandling ved krigsskader. Gjennom de siste årtier er metadon blitt det mest anvendte medikament i substitusjonsbehandling ved opiatavhengighet. Senere forskning har vist at metadon påvirker hjerterytmen. En studie har avdekket forlenget QTc-tid på minst 500 ms hos 16,2 % av pasienter som bruker metadon. En randomisert kontrollert sammenligningsstudie av metadon, levometadyl hydroklorid acetat (LAAM) og buprenorfin, har vist at metadon og LAAM gir signifikant forlenget QTc-tid, dvs. >470 ms hos menn og >490 ms hos kvinner, eller en forlengelse på minst 60 ms fra basislinjen. Det ser ut til å være doseavhengig forhold mellom metadon og QTc-tid. En norsk studie kartla forekomsten av forlenget QTc-tid hos pasienter i Legemiddelassistert rehabilitering (LAR) i Oslo. QTc-tiden ble sett i sammenheng med medikamenttype (metadon eller buprenorfin), dose, kjønn og behandlingens varighet. Studiet viste en forlengelse av QTc-tid til omkring 500 ms hos4,6% av pasientene som ble behandlet med metadon. Forlenget QTc-tid er forbundet med ventrikulære arytmier "Torsades de Pointes" og plutselig hjertestans. Den underliggende mekanismen skyldes blokkering av kalium-strømmen gjennom hjertets ionekanaler (human "ether-a-go-go-related" gene (hERG)).

Tilnærmet 50% dvs nær 3.000 av norske LAR-pasienter behandles med rasemisk metadon eller (R,S)-metadon. Metadonets stabiliserende virkning knyttes til R-metadon, mens S-metadonen blir betraktet som inaktiv. Både (R-) og (S)-metadon hemmer hERG-kanalen, men S-metadon binder til kanalen og hemmer utadrettet kalium-strøm i hjertemuskelceller ved lavere konsentrasjon enn (R)-metadon.

Formålet med denne studien er å kartlegge endringer i QTc-tid ved overgang fra (R,S)-metadon til R-metadon hos LAR-pasienter med kjent forlenget QTc-tid.

Hypotesen er at medikamentskifte fra (R,S)-metadon til (R)-metadon medfører en reduksjon i QTc-tid. Behandling med (R)-metadon kan være et viktig bidrag til pasienter som får forlenget QTc-tid ved bruk av racemisk metadon og som av ulike grunner ikke vil skifte til buprenorfin.

# Design, materiale, metoder og etiske betenkeligheter:

**Design:** Dette er en deskriptiv og prospektiv studie av pasient-kasuistikker.

Materiale: Femten LAR-pasienter med forlenget QTc-tid ved Oslo Universitetssykehus.

#### Inklusjonskriterier:

- Stabilisert på fast metadondose
- Fri for bruk av andre rusmidler
- Påvist forlengelse av hjertets ledningstid (QTc-tid), verdi over 500 mS.
- Alder 18 år eller eldre
- Signert skiftlig informert samtykke

## Eksklusjonskriterier:

- Problemer med fremmøte til daglige observerte inntak
- Alvorlige psykiatriske diagnoser eller ubehandlede alvorlige somatiske sykdommer, hvor symptomene og medisinering kan komplisere tolkningen av testresultatene
- Graviditet

**Metode:** Hjerterytmen vil bli studert med med 12-lednings-EKG. Serumnivået på metadon og elektrolytter vil bli målt henholdsvis før (Cmin) og 2-3 timer etter medikamentinntak (Cmaks). Videre vil det bli rusmiddelanalyse av spytt eller urin. Det vil bli skreenet for genetiske varianter.

Kliniske undersøkelser innbefatter registrering av henholdsvis subjektive og objektive abstinenssymptomer ved bruk av validerte spørreskjema - Subjective Opioid Withdrawal Symptoms (OOWS) og Objective Opioid Withdrawal Symptoms (SOWS).

**Betraktninger:** LAR-pasienter vil bli overført til daglige overvåkede inntak minst fem dager før skifte til (R)-metadon. R-metadon er tilgjengelig fra Tyskland under preparatnavnet L-Polamydon. Konverteringsforholdet vil være lik halvparten av stabilisert dose (eksempel 90 mg (R,S)-metadon vil erstattes med 45 mg L-Polamydon). Det er beregnet minst 10 dager mellom seponering av R,S (dag 8) og målingene for R-metadon (dag 18) for å tilfredsstille at S-metadonfraksjonen av (R,S)-metadon er eliminert (>10 halveringstider siden siste inntak) og at R-metadon ser stabilisert (>5 halveringstider for R-metadon).

Dag 1-5: Daglige overvåkede inntak av metadon på apotek eller tilsvarende Dag 8: Oppmøte på Oslo Universitetssykehus

Oppmøte på Oslo UniversitetssykehusFør medikamentinntak: Utfylling av spøl

- Før medikamentinntak: Utfylling av spørreskjema for kartlegging av abstinenssymptomer, EKG og blodprøver\* (herunder Cmin for metadon) (se avsnitt Blodprøver under) Urinprøve til Rusmiddelanalyse
- Seponere (R,S)-metadon og starte med (R)-metadon (L-Polamydon), halv dose av opprinnelige metadondose
- 2-3 timer etter medikamentinntak: Ny utfylling av spørreskjema for kartlegging av abstinenssymptomer, med blodprøver (herunder Cmaks for metadon se avsnitt Blodprøver under) og EKG

Dag 9-17: Daglige overvåkede inntak av L-Polamydon på apotek eller tilsvarende Dag 18 Oppmøte på Oslo Universitetssykehus

- Før medikamentinntak: Utfylling av spørreskjema for kartlegging av abstinenssymptomer, EKG og blodprøver\* (herunder Cmin for metadon)
- To-tre timer etter medikamentinntak: Ny utfylling av spørreskjema for kartlegging av abstinenssymptomer med blodprøver\* og EKG

### \*Blodprøver

- Elektrolytter (Na, Ca, Mg, K), TSH, fritt T4, kreatinin, estimert GFR, cystatin C, urea, ALAT, INR, troponin-T, CRP, differentialtelling av hvite blodlegemer tas før medikamentinntak dag 8 og 18
- Genetiske undersøkelser omfatter CYP screening (CYP3A4, CYP3A5, CYP2B6, CYP2D6, CYP2C9, CYP2C19, CYP3A4 med genotype for "long QT-time syndrome" og skreening for eventuelle polymorfisme for mu-receptor tas dag 8.
- Serum-metadon med enatiomerbestemmelse tas dag 8 og 18, henholdsvis før medikamentinntak (Cmin) og 2-3 timer etter medikamentinntak (Cmaks)
- Urinprøve til Rusmiddelanalyse tas dag 8 og 18

**Etiske betraktninger**: Pasienten vil motta muntlig og skriftlig informasjon om studiet. Deltakelse forutsetter skriftlig samtykke. Studiet inkluderer blodprøvetaking, EKG og klinisk undersøkelse med hensyn til subjektive og objektive abstinenssymptomer. Ingen av undersøkelsene regnes å innebære noe risiko for pasienten. Dersom undersøkelsen avdekker en signifikant reduksjon av pasientens QTc-tid, vil pasienten få tilbud om videre behandling med R-metadon (L-Polamydon).

**Statistiske betraktninger:** Studien vil omfatte alle LAR-pasienter i Oslo med kjent forlenget QTc-tid (korrigert QT-tid over 500 ms). Hver pasient vil være sin egen kontroll der positiv effekt defineres som reduksjon i korrigert QT-tid i forhold til patologisk utgangsverdi.

**Organisering:** Studiet vil være et samarbeidsprosjekt mellom følgende avdelinger ved Oslo universitetssykehus:

- Senter rus og avhengighet, Klinikk psykisk helse og avhengighet ved Dr. med. Peter Krajci
- Senter for rus og avhengighetsforskning (SERAF) ved professor emeritus Helge Waal
- Avdeling for farmakologi, Klinikk for diagnostikk og intervensjon ved dr med Mimi Stokke Opdal og professor dr med Odd Brørs
- Hjertemedisinsk avdeling, Medisinsk klinikk ved professor dr med Knut Gjesdal

#### Referanseliste

Waal H, Clausen T, Håseth A, Lillevold PH. SERAF RAPPORT 1/2010 Siste år med gamle retningslinjer Statusrapport 2009. Oslo: Senter for rus- og avhengighetsforskning; 2010

Anchersen K, Clausen T, Gossop M, Hansteen V, Waal H. Prevalence and clinical relevance of corrected QT interval prolongation during methadone and buprenorphine treatment: a mortality assessment study. Addiction 2009 Jun;104(6):993-9

Katchman AN, McGroary KA, Kilborn MJ, Kornick CA, Manfredi PL, Woosley RL, et al. Influence of opioid agonists on cardiac human ether-a-go-go-related gene K(+) currents. J Pharmacol Exp Ther 2002 Nov;303(2):688-94

Peles E, Bodner G, Kreek MJ, Rados V, Adelson M. Corrected-QT intervals as related to methadone dose and serum level in methadone maintenance treatment (MMT) patients: a cross-sectional study. Addiction 2007 Feb;102(2):289-300

Totah RA, Allen KE, Sheffels P, Whittington D, Kharasch ED. Enantiomeric metabolic interactions and stereoselective human methadone metabolism. J Pharmacol Exp Ther 2007 Apr;321(1):389-99

Charuvastra VC, Ouren J. Renal failure and treatment of a methadone maintenance patient. Med J Aust 1977 Sep 24;2(13):433-4

Handelsman L, Cochrane KJ, Aronson MJ, Ness R, Rubinstein KJ, Kanof PD. Two new rating scales for opiate withdrawal. Am J Drug Alcohol Abuse 1987;13(3):293-308